CLINICAL TRIAL: NCT07205783
Title: Open Radical Prostatectomy for Treatment of Organ Confined Prostate Cancer (Tumor Control and Functional Outcome)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Khalaf Elsayed, assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-9-2MD
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
Keywords: open radical prostatectomy prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cancer prostate (Experimental)
  Interventions: Procedure: open radical prostatectomy

INTERVENTIONS:
Procedure: open radical prostatectomy — open surgery to remove prostate gland and the tumor

SUMMARY:
In the last few decades not only the diagnosis but also the treatment options for prostate cancer have changed significantly. During this time the surgical procedure of open radical prostatectomy was substantially modified(1,2) and is nowadays considered a safe procedure providing high cancer control rates with low morbidity.(3) The main goal of radical prostatectomy regardless of the approach remains the eradication of cancer while preserving pelvic organ function,whenever possible.(4)

ELIGIBILITY:
Inclusion Criteria:

* Cancer prostate: confirmed by prostate biopsy Cancer stage: T2,T3

Exclusion Criteria:

* coagulopathy. Pulmonary diseases metastatic tumor

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 20 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2026-09-14 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
tumor control | 6 months
  percentage of tumor recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No